CLINICAL TRIAL: NCT04232787
Title: Discovering the Genetic Causes of Brugada Syndrome in Thais and Southeast Asian Population
Brief Title: Southeast Asian Brugada Syndrome Cohort
Acronym: SEA-BrS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: National Research Council of Thailand (Other Government); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Apichai Khongphatthanayothin, MD, Professor of Pediatrics, Division of Pediatric Cardiology, Department of Pediatrics, Faculty of Medicine, Chulalongkorn University
Other Study IDs: 2558-114
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Brugada Syndrome
Keywords: Brugada Syndrome; Genetics; Epidemiology; Thai; Southeast Asia
MeSH Terms: conditions — Brugada Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Thai patients with diagnosed Brugada syndrome by confirmed Brugada type 1 ECG.
- Control: Healthy volunteers without Brugada marker from ECG.

SUMMARY:
Brugada syndrome (BrS) is the leading cause of sudden death in young Asian adults including Thailand. This syndrome may be hereditary and involve mutations in certain genes. Aim of the study is to identify the relationship between genetic variants and the diagnosis/clinical severity of patients with BrS.

DETAILED DESCRIPTION:
This cohort study recruits BrS patients with confirmed Brugada type 1 ECG and healthy volunteers in Thailand. Data collection consists of demographic, clinical data, ECG and blood sample for genetic studies. Genotyping was done by whole genome sequencing and SNP array then compared between cases and controls. Each BrS patient will be followed up prospectively for symptoms and AICD shock. Subsequently, the study will analyze relationship between genetic variants and clinical data against clinical severity of BrS patients.

ELIGIBILITY:
Inclusion Criteria:

* Thai nationality
* The patient has at least one of confirmed Brugada type 1 ECG in at least one of right precordial leads (v1 or v2) with or without pharmacologic provocative testing. The confirmed ECG is standard 12 lead ECG or Brugada lead

Exclusion Criteria:

* The patient has other cardiac diseases such as ischemic heart disease, valvular heart disease, congenital heart disease, myocarditis and pericarditis
* The patient has type 2 or type 3 Brugada ECG without type 1 ECG during pharmacologic provocative testing and/or Brugada lead
* The patient had one time of Brugada type 1 ECG during drug use without reproducibility

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Thai Brugada syndrome patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2016-01-28 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between genetic variants and Brugada syndrome (Brugada syndrome phenotype) | 7 years
  Case-Control study of genetic variants in BrS cases vs controls. Genetic study was done by whole genome sequencing and SNP array. Association analysis assessed by polygenic risk score and regression coefficients.

SECONDARY OUTCOMES:
Natural history of Brugada syndrome (survival from arrhythmic events) | 7 years
  Cohort study to followed up BrS patients with or with arrhythmic events which assessed by survival curve analysis.
Epidemiology of Brugada syndrome | 7 years
  To study prevalence of Brugada syndrome in Thailand.

CONTACTS AND LOCATIONS:
Overall Officials: Koonlawee Nademanee, MD, Study Chair — Chulalongkorn University; Yong Poovorawan, MD, Study Director — Chulalongkorn University; Apichai Khongphatthanayothin, MD, Principal Investigator — Chulalongkorn University
Locations (11):
- Thailand (11):
  - Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok
  - Vajira Hospital, Dusit, Bangkok
  - Chulalongkorn University, Pathum Wan, Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok
  - Bhumibol Adulyadej RTAF Hospital, Sai Mai, Bangkok
  - Bumrungrad International Hospital, Vadhana, Bangkok
  - Pacific Rim Electrophysiology Research Institute Data Coordinating Center, Vadhana, Bangkok
  - Bangkok Hospital, Bangkok
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Queen Sirikit Heart Center of the Northeast, Khon Kaen
  - Central Chest Hospital, Nonthaburi

IPD SHARING:
Plan to Share IPD: Yes
Medical journals, abstract submissions and results database

REFERENCES:
- [Result] Deo R, Albert CM. Epidemiology and genetics of sudden cardiac death. Circulation. 2012 Jan 31;125(4):620-37. doi: 10.1161/CIRCULATIONAHA.111.023838. No abstract available. PMID 22294707
- [Result] Priori SG, Wilde AA, Horie M, Cho Y, Behr ER, Berul C, Blom N, Brugada J, Chiang CE, Huikuri H, Kannankeril P, Krahn A, Leenhardt A, Moss A, Schwartz PJ, Shimizu W, Tomaselli G, Tracy C. HRS/EHRA/APHRS expert consensus statement on the diagnosis and management of patients with inherited primary arrhythmia syndromes: document endorsed by HRS, EHRA, and APHRS in May 2013 and by ACCF, AHA, PACES, and AEPC in June 2013. Heart Rhythm. 2013 Dec;10(12):1932-63. doi: 10.1016/j.hrthm.2013.05.014. Epub 2013 Aug 30. No abstract available. PMID 24011539
- [Result] Nademanee K, Veerakul G, Nimmannit S, Chaowakul V, Bhuripanyo K, Likittanasombat K, Tunsanga K, Kuasirikul S, Malasit P, Tansupasawadikul S, Tatsanavivat P. Arrhythmogenic marker for the sudden unexplained death syndrome in Thai men. Circulation. 1997 Oct 21;96(8):2595-600. doi: 10.1161/01.cir.96.8.2595. PMID 9355899
- [Result] Bezzina CR, Barc J, Mizusawa Y, Remme CA, Gourraud JB, Simonet F, Verkerk AO, Schwartz PJ, Crotti L, Dagradi F, Guicheney P, Fressart V, Leenhardt A, Antzelevitch C, Bartkowiak S, Borggrefe M, Schimpf R, Schulze-Bahr E, Zumhagen S, Behr ER, Bastiaenen R, Tfelt-Hansen J, Olesen MS, Kaab S, Beckmann BM, Weeke P, Watanabe H, Endo N, Minamino T, Horie M, Ohno S, Hasegawa K, Makita N, Nogami A, Shimizu W, Aiba T, Froguel P, Balkau B, Lantieri O, Torchio M, Wiese C, Weber D, Wolswinkel R, Coronel R, Boukens BJ, Bezieau S, Charpentier E, Chatel S, Despres A, Gros F, Kyndt F, Lecointe S, Lindenbaum P, Portero V, Violleau J, Gessler M, Tan HL, Roden DM, Christoffels VM, Le Marec H, Wilde AA, Probst V, Schott JJ, Dina C, Redon R. Common variants at SCN5A-SCN10A and HEY2 are associated with Brugada syndrome, a rare disease with high risk of sudden cardiac death. Nat Genet. 2013 Sep;45(9):1044-9. doi: 10.1038/ng.2712. Epub 2013 Jul 21. PMID 23872634
- [Derived] Chimparlee N, Prechawat S, Khongphatthanayothin A, Mauleekoonphairoj J, Lekchuensakul S, Wongcharoen W, Makarawate P, Sahasatas D, Krittayaphong R, Amnueypol M, Anannab A, Ngarmukos T, Vardhanabhuti S, Sutjaporn B, Wandee P, Veerakul G, Bezzina CR, Poovorawan Y, Nademanee K. Clinical Characteristics of SCN5A p.R965C Carriers: A Common Founder Variant Predisposing to Brugada Syndrome in Thailand. Circ Genom Precis Med. 2021 Jun;14(3):e003229. doi: 10.1161/CIRCGEN.120.003229. Epub 2021 Jun 7. No abstract available. PMID 34092119
- [Derived] Makarawate P, Glinge C, Khongphatthanayothin A, Walsh R, Mauleekoonphairoj J, Amnueypol M, Prechawat S, Wongcharoen W, Krittayaphong R, Anannab A, Lichtner P, Meitinger T, Tjong FVY, Lieve KVV, Amin AS, Sahasatas D, Ngarmukos T, Wichadakul D, Payungporn S, Sutjaporn B, Wandee P, Poovorawan Y, Tfelt-Hansen J, Tanck MWT, Tadros R, Wilde AAM, Bezzina CR, Veerakul G, Nademanee K. Common and rare susceptibility genetic variants predisposing to Brugada syndrome in Thailand. Heart Rhythm. 2020 Dec;17(12):2145-2153. doi: 10.1016/j.hrthm.2020.06.027. Epub 2020 Jun 30. PMID 32619740
- See also: Project database — https://redcap.prepdb.org/index.php?action=myprojects